CLINICAL TRIAL: NCT04714073
Title: Effect of Itraconazole on the Pharmacokinetics of a Single Oral Dose of BI 706321 in Healthy Male Subjects (an Open-label, Two-period Fixed Sequence Design Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 706321 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1425-0010; 2020-004388-22 (EudraCT Number)
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: In the first treatment period all subjects are planned to undergo the reference treatment (R), and in the second treatment period all subjects are planned to undergo the test treatment (T).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 706321 (Reference (R))/ BI 706321 + Itraconazole (Test (T)) (Experimental): On trial day 1 of treatment period 1, a single oral dose of 1 film-coated tablet of 2 milligram (mg) BI 706321 was administered with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment (R).
  In treatment period 2: 200 mg itraconazole was administered as an oral solution formulation (concentration: 20 mL of 10 mg/mL) once daily for 14 days orally with 240 mL of water after an overnight fast of at least 9 h, starting from day -3 up to day 11 of period 2. On day 1 of period 2 (1 h after the itraconazole administration) a single oral dose of 1 film-coated tablet of 2 mg BI 706321 was administered with 240 mL of water after an overnight fast of at least 10 h (Test Treatment (T)).
  There was a washout interval of at least 14 days between the administrations of BI 706321 in the 2 trial periods.
  Interventions: Drug: BI 706321; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 706321 — Treatment period 1: Single oral dose of 1 film-coated tablet administered with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) Treatment period 2: On day 1 of period 2 (1 h after the itraconazole administration) a single oral dose of 1 film-coated tablet administered with 240 mL of water after an overnight fast of at least 10 h.
Drug: Itraconazole — Treatment period 2: Administered as an oral solution formulation once daily for 14 days orally with 240 mL of water after an overnight fast of at least 9 h, starting from day -3 up to day 11 of period 2.

SUMMARY:
To investigate the pharmacokinetics of a single oral dose of BI 706321 when given alone or in combination with itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (body temperature, blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Effect of itraconazole on the pharmacokinetics of a single oral dose of BI 706321 in healthy male subjects (an open-label, two-period fixed sequence design study)
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 706321 (R)/ BI 706321 + Itraconazole (T): On trial day 1 of treatment period 1, a single oral dose of 1 film-coated tablet of 2 milligram (mg) BI 706321 was administered with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment (R).
  In treatment period 2: 200 mg itraconazole was administered as an oral solution formulation (concentration: 20 mL of 10 mg/mL) once daily for 14 days orally with 240 mL of water after an overnight fast of at least 9 h, starting from day -3 up to day 11 of period 2. On day 1 of period 2(1 h after the itraconazole administration) a single oral dose of 1 film-coated tablet of 2 mg BI 706321 was administered with 240 mL of water after an overnight fast of at least 10 h (Test Treatment (T)).
  There was a washout interval of at least 14 days between the administrations of BI 706321 in the 2 trial periods.
Period: Period 1 (+Washout Period)
Arm/Group | BI 706321 (R)/ BI 706321 + Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0
Period: Period 2
Arm/Group | BI 706321 (R)/ BI 706321 + Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were treated with at least 1 dose of study drug.
Arm/Group | BI 706321 (R)/ BI 706321 + Itraconazole (T)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 706321 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 706321 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours (h) (1h for period 2) before and at 0.5h to 190h after BI 706321 administration in each period. Further at 214h to 550h after BI 706321 administration in period 2.
Population: Pharmacokinetic parameter analysis set (PKS): All subjects in the treated set who provided at least 1 Pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: Hours * nanomoles / liter
Groups:
- BI 706321 Alone (Reference Treatment (R)): On trial day 1 of treatment period 1, a single oral dose of 1 film-coated tablet of 2 milligram (mg) BI 706321 was administered with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment (R).
- BI 706321 + Itraconazole (Test Treatment(T)): In treatment period 2: 200 mg itraconazole was administered as an oral solution formulation (concentration: 20 mL of 10 mg/mL) once daily for 14 days orally with 240 mL of water after an overnight fast of at least 9 h, starting from day -3 up to day 11 of period 2. On day 1 of period 2(1 h after the itraconazole administration) a single oral dose of 1 film-coated tablet of 2 mg BI 706321 was administered with 240 mL of water after an overnight fast of at least 10 h (Test Treatment (T)).
Arm/Group | BI 706321 Alone (Reference Treatment (R)) | BI 706321 + Itraconazole (Test Treatment(T))
Number analyzed (Participants) | 14 | 14
Hours * nanomoles / liter | 60.99 (NA) — Adjusted geometric standard error = 1.10 | 133.45 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: BI 706321 Alone (Reference Treatment (R)) vs BI 706321 + Itraconazole (Test Treatment(T)); The statistical model used for the analysis of the primary PK endpoints was an analysis of variance (ANOVA) model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'subjects' and 'treatment'. The effect 'subject' was considered as random, whereas 'treatment' was considered as fixed; Test type: Other; Ratio of geometric means (%) = 218.81, 90% CI 2-sided [194.06 to 246.72] — The estimated parameter was the adjusted geometric mean ratio (%): BI 706321 + Itraconazole (Test Treatment(T))/BI 706321 alone (Reference Treatment (R)). Intra-individual geometric coefficient of variation (gCV) [%] = 18.1

2. Primary Outcome: Maximum Measured Concentration of BI 706321 in Plasma (Cmax)
Description: Maximum measured concentration of BI 706321 in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomoles / liter
Arm/Group | BI 706321 Alone (Reference Treatment (R)) | BI 706321 + Itraconazole (Test Treatment(T))
Number analyzed (Participants) | 14 | 14
nanomoles / liter | 2.22 (NA) — Adjusted geometric standard error = 1.14 | 3.47 (NA) — Adjusted geometric standard error = 1.14
Statistical Analysis 1: Comparison: BI 706321 Alone (Reference Treatment (R)) vs BI 706321 + Itraconazole (Test Treatment(T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (%) = 156.29, 90% CI 2-sided [135.04 to 180.89] — The estimated parameter was the adjusted geometric mean ratio (%): BI 706321 + Itraconazole (Test Treatment(T))/BI 706321 alone (Reference Treatment (R)). Intra-individual geometric coefficient of variation (gCV) [%] = 22.1

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 706321 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 706321 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: Hours * nanomoles / liter
Arm/Group | BI 706321 Alone (Reference Treatment (R)) | BI 706321 + Itraconazole (Test Treatment(T))
Number analyzed (Participants) | 14 | 14
Hours * nanomoles / liter | 50.89 (NA) — Adjusted geometric standard error = 1.12 | 113.54 (NA) — Adjusted geometric standard error = 1.12
Statistical Analysis 1: Comparison: BI 706321 Alone (Reference Treatment (R)) vs BI 706321 + Itraconazole (Test Treatment(T)); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (%) = 223.12, 90% CI 2-sided [198.61 to 250.66] — The estimated parameter was the adjusted geometric mean ratio (%): BI 706321 + Itraconazole (Test Treatment(T))/BI 706321 alone (Reference Treatment (R)). Intra-individual geometric coefficient of variation (gCV) [%] = 17.5

ADVERSE EVENTS:
Time Frame: BI 706321 (BI) in period (p) 1: From BI administration in p1 until 8 days (d) thereafter, up to 8d. Itraconazole (Itra) alone in p2: From 1st Itra administration in p2 until BI administration in p2 or until last Itra administration in p2 if discontinuation prior to BI administration in p2 + 8d, up to 11d. BI+Itra in period 2: From BI administration in p2 until 8d after last study drug administration, up to 18d. Continues in description.
Description: Continuation of time frames:
  Total BI: From BI administration in p1 until 8d thereafter and from BI administration in p2 until 8d after last study drug administration, up to 26d.
  Total: From BI administration in p1 until 8d after last study drug administration in p2, up to 29d.
  Safety analyses were based on the treated set (TS). The TS included all subjects who were treated with at least 1 dose of study drug.
Groups:
- BI 706321 in Period 1: On trial day 1 of treatment period 1, a single oral dose of 1 film-coated tablet of 2 milligram (mg) BI 706321 was administered with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) as reference treatment (R).
- Itraconazole Alone in Period 2: In treatment period 2: 200 mg itraconazole was administered as an oral solution formulation (concentration: 20 mL of 10 mg/mL) once daily orally with 240 mL of water after an overnight fast of at least 9 h, starting from day -3 up to day 1 of period 2.
- BI 706321+Itraconazole in Period 2: 200 milligrams (mg) itraconazole were administered as oral solution formulation (concentration: 20 mL of 10 mg/milliliter (mL)) once daily with 240 mL of water after an overnight fast of at least 9 hours (h), starting from day 1 up to day 11 of period 2. On day 1 of period 2(1 h after the itraconazole administration) a single oral dose of 1 film-coated tablet of 2 mg BI 706321 was administered with 240 mL of water after an overnight fast of at least 10 h.
- Total BI 706321: A total over all on treatment phase involving BI 706321.
- Total: A total over all on treatment phase included in this analysis.
Arm/Group | BI 706321 in Period 1 | Itraconazole Alone in Period 2 | BI 706321+Itraconazole in Period 2 | Total BI 706321 | Total
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 3/14 | 5/14 | 8/14 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 706321 in Period 1 (N=14) | Itraconazole Alone in Period 2 (N=14) | BI 706321+Itraconazole in Period 2 (N=14) | Total BI 706321 (N=14) | Total (N=14)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 3 | 5
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 4 | 0 | 1 | 4 | 4
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review Prior to any Submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI´s intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04714073/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT04714073/SAP_001.pdf